CLINICAL TRIAL: NCT01988493
Title: A Multicenter, Randomized, Phase Ib/II Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of MSC2156119J as Monotherapy Versus Sorafenib in Asian Subjects With MET+ Advanced Hepatocellular Carcinoma and Child-Pugh Class A Liver Function
Brief Title: Efficacy, Safety, and Pharmacokinetic of MSC2156119J in Asian Participants With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200095-004
Record Dates: First submitted 2013-11-01; First posted 2013-11-20 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular; MSC2156119J; Sorafenib; Recommended Phase 2 dose
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tepotinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1b: Tepotinib 300 mg (Experimental): Participants received Tepotinib 300 milligram (mg) orally once daily over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Interventions: Drug: Tepotinib 300 mg
- Phase 1b: Tepotinib 500 mg (Experimental): Participants received Tepotinib 500 mg orally once daily over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Interventions: Drug: Tepotinib 500 mg
- Phase 1b: Tepotinib 1000 mg (Experimental): Participants received Tepotinib 1000 mg orally once daily over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Interventions: Drug: Tepotinib 1000 mg
- Phase 2: Tepotinib (Experimental): Participants randomized to receive Tepotinib recommended Phase 2 dose (RP2D) determined from Phase 1b over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Interventions: Drug: Tepotinib
- Phase 2 Sorafenib (Experimental): Participants randomized to receive Sorafenib 400 mg orally twice daily over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Tepotinib 300 mg — Participants received Tepotinib 300 milligram (mg) orally once daily over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Arms: Phase 1b: Tepotinib 300 mg
Drug: Tepotinib 500 mg — Participants received Tepotinib 500 mg orally once daily over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Arms: Phase 1b: Tepotinib 500 mg
Drug: Tepotinib 1000 mg — Participants received Tepotinib 1000 mg orally once daily over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal
  Arms: Phase 1b: Tepotinib 1000 mg
Drug: Tepotinib — Participants randomized to receive Tepotinib recommended Phase 2 dose (RP2D) determined from Phase 1b over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Arms: Phase 2: Tepotinib
Drug: Sorafenib — Participants randomized to receive Sorafenib 400 mg orally twice daily over a 21-day cycle until disease progression, intolerable toxicity or participant withdrawal.
  Arms: Phase 2 Sorafenib

SUMMARY:
This is an open-label, integrated, Phase 1b/2 trial to determine the recommended Phase 2 dose (RP2D) and to evaluate the efficacy, safety, and pharmacokinetic of MSC2156119J as first-line treatment versus sorafenib in subjects with MET+, Barcelona Clinic Liver Cancer (BCLC) Stage C, systemic treatment naive advanced hepatocellular carcinoma (HCC) and Child-Pugh class A liver function.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HCC
* Participants were either intermediate HCC of BCLC Stage B, who were not eligible for surgical and/or local-regional therapies or who had progressive disease (PD) after surgical and/or local-regional therapies (note: the local-regional therapy must not contain sorafenib), or advanced HCC of BCLC Stage C
* Participants who had disease progression on or were intolerant to the prior standard treatment for advanced HCC (phase Ib Korean subjects only)
* A tumor biopsy was required for determining MET status
* MET+ status (Phase 2 only), as determined by the central laboratory (Phase 1b retrospectively, Phase 2 for participant selection) were defined in the protocol
* Child-Pugh class A with no encephalopathy according to the screening assessment
* Asian male or female, 18 years of age or older
* Measurable disease in accordance with RECIST v1.1 (Phase 2 only)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2
* Eligible for treatment with sorafenib, was assessed by investigators according to the Package Insert and clinical judgment (Phase 2 only)
* Signed and dated informed consent indicating that the participants had been informed of all the pertinent aspects of the trial prior to enrollment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures
* Life expectancy was judged by the investigator of at least 3 months

Exclusion Criteria:

* Prior systemic anticancer treatment for advanced HCC, included targeted therapy (for example, sorafenib), chemotherapy, or any other investigational agent (Phase 2 only)
* Prior treatment with any agent targeting the hepatocyte growth factor (HGF)/c-Met pathway
* Prior local-regional therapy within 4 weeks prior to Day 1 of trial treatment
* Prior history of liver transplant
* Laboratory index at baseline were defined in the protocol
* Past or current history of neoplasm other than HCC, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer curatively treated and with no evidence of disease for at least 5 years
* Known central nervous system (CNS) or brain metastasis that is either symptomatic or untreated
* Medical history of difficulty swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested products
* Clinically significant gastrointestinal bleeding within 4 weeks before trial entry
* Peripheral neuropathy Grade greater than or equal to 2 (Common Terminology Criteria for Adverse Events [CTCAE] v4.0)
* Impaired cardiac function was defined in the protocol
* Hypertension uncontrolled by standard therapies
* Participants with a family history of long QT syndrome or who take any agent that is known to prolong QT/QTc interval
* Known human immunodeficiency virus (HIV) infection
* Particpants who had acute pancreatitis and/or chronic pancreatitis, with elevated lipase and/or amylase, clinical symptoms, and/or imaging studies that are indicative of the diagnosis (Mainland Chinese participants only)
* Known or suspected drug hypersensitivity to any ingredients of sorafenib (Phase 2 only) and MSC2156119J
* Female participants who were pregnant or lactating, or males and females of reproductive potential not willing or not able to employ a highly effective method of birth control/contraception to prevent pregnancy from 2 weeks before receiving study drug until 3 months after receiving the last dose of study drug
* Concurrent treatment with a non-permitted drug
* Substance abuse, other acute or chronic medical or psychiatric condition, or laboratory abnormalities that may increase the risk associated with trial participation in the opinion of the investigator
* Participation in another clinical trial within the past 28 days
* Previous anticancer treatment-related toxicities not recovered to baseline or Grade 0-1 (except alopecia and peripheral neuropathy)
* Participants with any concurrent medical condition or disease that will potentially compromise the conduct of the study at the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (43):
- China (15):
  - 307 Hosptial of PLA, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Area Command of Chinese PLA, Fuzhou, Fujian
  - Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Third Xiangya Hospital of Central South University, Changsha, Hu'nan
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shanghai Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Cancer Hospital, Tianjin Medical University, Tianjin, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Zhejiang, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing
- South Korea (18):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - National Cancer Center, Goyang-si
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Pusan National University Yangsan Hospital, Yangsan
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Liou Ying, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

REFERENCES:
- [Result] Ryoo BY, Cheng AL, Ren Z, Kim TY, Pan H, Rau KM, Choi HJ, Park JW, Kim JH, Yen CJ, Lim HY, Zhou D, Straub J, Scheele J, Berghoff K, Qin S. Randomised Phase 1b/2 trial of tepotinib vs sorafenib in Asian patients with advanced hepatocellular carcinoma with MET overexpression. Br J Cancer. 2021 Jul;125(2):200-208. doi: 10.1038/s41416-021-01380-3. Epub 2021 May 10. PMID 33972742
- [Derived] Xiong W, Hietala SF, Nyberg J, Papasouliotis O, Johne A, Berghoff K, Goteti K, Dong J, Girard P, Venkatakrishnan K, Strotmann R. Exposure-response analyses for the MET inhibitor tepotinib including patients in the pivotal VISION trial: support for dosage recommendations. Cancer Chemother Pharmacol. 2022 Jul;90(1):53-69. doi: 10.1007/s00280-022-04441-3. Epub 2022 Jun 30. PMID 35771259
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=200095-004
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled 06 Jan 2014. Last participant last visit: 03 Dec 2020.
Pre-assignment Details: A total of 27 participants were enrolled in Phase 1b part of the study and a total of 90 participants were enrolled in phase 2 part of the study. Participants enrolled in phase 1b were not eligible for randomization in phase 2.
Period: Overall Study
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg | Phase 2: Tepotinib | Phase 2 Sorafenib
Started | 7 | 14 | 6 | 45 | 45
Treated | 7 | 14 | 6 | 45 | 44
Safety Population | 7 | 14 | 6 | 45 | 44
Completed | 7 | 14 | 6 | 45 | 44
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who had received any dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg | Phase 2: Tepotinib | Phase 2 Sorafenib | Total
Number analyzed (Participants) | 7 | 14 | 6 | 45 | 44 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 11 | 5 | 34 | 37 | 93
  >=65 years | 1 | 3 | 1 | 11 | 7 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4 | 3 | 11
  Male | 6 | 12 | 5 | 41 | 41 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 14 | 6 | 45 | 44 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 14 | 6 | 45 | 44 | 116
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants Experiencing Dose Limiting Toxicity
Description: Dose limiting toxicity (DLT) was defined as toxicities at any dose level and judged to be related to the study treatment by investigator and/or the sponsor. DLTs included Grade 4 neutropenia for more than 7 days; Grade greater than or equal to (>=) 3 febrile neutropenia for more than 1 day; Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with non-traumatic bleeding; Grade >= 3 uncontrolled nausea/vomiting and/or diarrhea despite adequate and optimal treatment and Grade >= 3 any non-hematological adverse event (AE), except the aforementioned gastrointestinal events and alopecia. Number of participants who experienced DLT during phase 1b were reported.
Time Frame: Day 1 to Day 21 of Cycle 1 (each cycle is 21 days)
Population: Dose Limiting Toxicity (DLT) set included all participants who experienced a DLT during Cycle 1, or received at least 80 percent of all planned doses of treatment during Cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 6 | 12 | 5
Participants | 0 | 0 | 0

2. Primary Outcome: Phase 1b: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug and assessed up to 94 weeks. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 30 after the last dose of study treatment, assessed up to 94 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
Participants
  Any TEAE | 7 | 14 | 6
  Any Serious TEAE | 2 | 9 | 4

3. Primary Outcome: Phase 2: Time to Progression (TTP) Based on Tumor Assessment by an Independent Review Committee (IRC)
Description: TTP was defined as the time in months from randomization to date of the observation of radiological progressive disease (PD) (based on Response Evaluation Criteria in Solid Tumors [RECIST] v1.1) assessed by an IRC. PD is defined as at least 20 percent (%) increase in sum of diameters of target lesions, taking as reference as smallest sum on study; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must demonstrate an absolute increase of at least 5 millimeter (mm).
Time Frame: From randomization to date of the observation of radiological progressive disease, assessed up to maximum 3.8 years
Population: The modified intent-to treat (mITT) analysis set in the Phase 2 part of this study included all participants with Mesenchymal-epithelial transition (MET)+ hepatocelluar carcinoma (HCC) who were randomized to study treatment.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Months | 2.9 [2.7 to 5.3] | 1.4 [1.4 to 1.6]
Statistical Analysis 1: Comparison: Phase 2: Tepotinib vs Phase 2 Sorafenib; Test type: Equivalence — Sample size required 100 TTP events to ensure 80% power with a two-sided significance level of 10% for rejecting the null hypothesis of equal treatment effect between treatment arms; p = 0.0087, Log Rank; Hazard Ratio (HR) = 0.46, 90% CI 2-sided [0.28 to 0.76]

4. Secondary Outcome: Phase 2: Progression Free Survival (PFS) Time Based on Tumor Assessment by the Independent Review Committee (IRC)
Description: Progression-free survival (PFS) time was defined as the time in months from randomization to either first observation of disease progression (based on RECIST v1.1) or occurrence of death due to any cause within 84 days of either randomization or the last tumor assessment. PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 millimeter(mm). PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Up to 2.8 years
Population: The mITT analysis set in the Phase 2 part of this study included all participants with MET+ HCC who were randomized to study treatment.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Months | 2.8 [1.4 to 4.2] | 1.4 [1.4 to 1.6]
Statistical Analysis 1: Comparison: Phase 2: Tepotinib vs Phase 2 Sorafenib; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.0229, Log Rank; Hazard Ratio (HR) = 0.53, 90% CI [0.33 to 0.84]

5. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Overall survival time was measured as time in months between the date of randomization and the date of death.
Time Frame: Time from randomization to the date of death or up to 6.9 years
Population: as for outcome 4
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Months | 9.3 [5.9 to 17.9] | 8.6 [6.4 to 9.8]
Statistical Analysis 1: Comparison: Phase 2: Tepotinib vs Phase 2 Sorafenib; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.2333, Log Rank; Hazard Ratio (HR) = 0.71, 90% CI [0.45 to 1.14]

6. Secondary Outcome: Phase 2: Time to Progression (TTP) Based on Tumor Assessment by Investigator
Description: TTP was defined as the time in months from randomization to date of the observation of radiological PD (based on RECIST v1.1) assessed by the investigator. PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization to date of the observation of radiological progressive disease, assessed up to maximum 2.8 years
Population: as for outcome 4
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Months | 5.6 [3.0 to 7.6] | 2.8 [1.5 to 2.8]
Statistical Analysis 1: Comparison: Phase 2: Tepotinib vs Phase 2 Sorafenib; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.0059, Log Rank; Hazard Ratio (HR) = 0.45, 90% CI [0.28 to 0.73]

7. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-infinity) of Tepotinib
Description: The AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: The Pharmacokinetic (PK) analysis included all participants who had received at least 1 dose of Tepotinib and who had provided at least 1 plasma concentration measurement of Tepotinib after the first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
nanogram hour per milliliter (ng*h/mL)
  Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, AUC(0-inf) dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, AUC(0-inf) dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, AUC(0-inf) dependent on Lambda(z) were not determined.
  Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, AUC(0-inf) dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, AUC(0-inf) dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, AUC(0-inf) dependent on Lambda(z) were not determined.

8. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-t) of Tepotinib
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration is at or above the lower limit of quantification (LLLQ). AUC(0-t) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: The PK analysis set was used. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at each specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 5 | 14 | 6
ng*h/mL
  Day 1 of Cycle 1 | 4700 (12.1) | 6760 (28.0) | 11900 (40.3)
  Day 15 of Cycle 1: number analyzed (Participants) | 5 | 11 | 6
  Day 15 of Cycle 1 | 11800 (35.7) | 16700 (29.7) | 28600 (38.8)

9. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration-Time Curve Within 1 Dosing Interval (AUC 0-tau) of Tepotinib
Description: AUC (0-tau) is the area under the plasma concentration time curve within 1 dosing interval.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 5 | 14 | 6
ng*h/mL
  Day 1 of Cycle 1 | 4700 (12.1) | 6760 (28.0) | 11900 (40.3)
  Day 15 of Cycle 1: number analyzed (Participants) | 5 | 11 | 6
  Day 15 of Cycle 1 | 11800 (35.7) | 16700 (29.7) | 28600 (38.8)

10. Secondary Outcome: Phase 1b: Maximum Observed Plasma Concentration (Cmax) of Tepotinib
Description: Cmax is the maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: The PK analysis set was used. Here "Number Analyzed" signifies those participants who were evaluable for specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
ng/mL
  Day 1 of Cycle 1 | 266 (24.7) | 394 (30.4) | 680 (44.0)
  Day 15 of Cycle 1: number analyzed (Participants) | 6 | 12 | 6
  Day 15 of Cycle 1 | 585 (30.8) | 815 (31.6) | 1370 (36.3)

11. Secondary Outcome: Phase 1b: Minimum Observed Plasma Concentration (Cmin) of Tepotinib
Description: Cmin is minimum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 15 of Cycle 1 (each Cycle is 21 days)
Population: The PK analysis set was used. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 5 | 11 | 6
ng/mL | 398 (39.0) | 529 (43.6) | 1010 (38.8)

12. Secondary Outcome: Phase 1b: Average Observed Plasma Concentration (Cav) of Tepotinib
Description: Cavg is the average plasma concentration within 1 dosing interval obtained directly from the concentration versus time curve.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 5 | 11 | 6
ng/mL | 494 (35.7) | 696 (29.7) | 1190 (38.8)

13. Secondary Outcome: Phase 1b: Time to Reach Maximum Plasma Concentration (Tmax) of Tepotinib
Description: Tmax is time to reach maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
Hours
  Day 1 of Cycle 1 | 8.00 [4.00 to 10.00] | 8.00 [4.00 to 24.00] | 10.00 [8.00 to 10.00]
  Day 15 of Cycle 1: number analyzed (Participants) | 6 | 12 | 6
  Day 15 of Cycle 1 | 6.00 [0.25 to 8.03] | 8.00 [0.25 to 10.00] | 8.00 [0.00 to 10.00]

14. Secondary Outcome: Phase 1b: Apparent Volume of Distribution During the Terminal Phase (Vz/f) of Tepotinib
Description: The Vz/f was defined as the theoretical volume in which the total amount of required to uniformly distribute to produce the desired plasma concentration. Apparent volume of distribution after oral dose (Vz/F) was influenced by the fraction absorbed. The Vz/f was calculated by dividing the dose with area under the concentration time curve from time zero to infinity multiplied with terminal elimination rate constant Lambda(z). Vz/f=Dose/AUC(0-inf)* Lambda(z).
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: The PK analysis included all participants who had received at least 1 dose of Tepotinib and who had provided at least 1 plasma concentration measurement of Tepotinib after the first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
Liter
  Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z) , Therefore, Vz/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z) , Therefore, Vz/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z) , Therefore, Vz/f dependent on Lambda(z) were not determined.
  Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Vz/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Vz/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Vz/f dependent on Lambda(z) were not determined.

15. Secondary Outcome: Phase 1b: Apparent Total Body Clearance From Plasma (CL/f) of Tepotinib
Description: The CL/f is a measure of the rate at which it was metabolized or eliminated by normal biological processes. Clearance obtained after oral dose was influenced by the fraction of the dose absorbed. The CL/F from plasma was calculated using the formula: Dose divided by area under the concentration time curve from time zero to infinity (AUC0-inf).
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
liter per hour (L/h)
  Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, CL/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, CL/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, CL/f dependent on Lambda(z) were not determined.
  Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, CL/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, CL/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, CL/f dependent on Lambda(z) were not determined.

16. Secondary Outcome: Phase 1b: Apparent Volume of Distribution During the Steady State (Vss/f) of Tepotinib
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss/f after oral dose was influenced by the fraction absorbed.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
liter
  Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z).Therefore, Vss/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z).Therefore, Vss/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z).Therefore, Vss/f dependent on Lambda(z) were not determined.
  Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z).Therefore, Vss/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z).Therefore, Vss/f dependent on Lambda(z) were not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z).Therefore, Vss/f dependent on Lambda(z) were not determined.

17. Secondary Outcome: Phase 1b: Apparent Terminal Elimination Rate Constant Lambda(z) of Tepotinib
Description: Lambda(z) was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1 per hour
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
1 per hour
  Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Lambda(z) was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Lambda(z) was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Lambda(z) was not determined.
  Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Lambda(z) was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Lambda(z) was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, Lambda(z) was not determined.

18. Secondary Outcome: Phase 1b: Apparent Terminal Half-life (t1/2) of Tepotinib
Description: Apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours postdose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg
Number analyzed (Participants) | 7 | 14 | 6
Hours
  Day 1 | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, t1/2 dependent on Lambda Z were not determined. | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, t1/2 dependent on Lambda Z were not determined. | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, t1/2 dependent on Lambda Z were not determined.
  Day 15 | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, t1/2 dependent on Lambda Z were not determined. | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, t1/2 dependent on Lambda Z were not determined. | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant Lambda(z). Therefore, t1/2 dependent on Lambda Z were not determined.

19. Secondary Outcome: Phase 2: Time-to-Symptomatic Progression (TTSP)
Description: Time-to-symptomatic progression was defined as time (in months) from first study drug administration to the date of deterioration of symptoms assessed by Functional Assessment of Cancer Therapy Hepatobiliary Symptom Index 8 (FHSI-8) (defined as at least a 4-point increase, i.e., higher score, compared with baseline value), or deterioration to Eastern Cooperative Oncology Group (ECOG) performance score 4, or death. FHSI-8 assesses hepatobiliary cancer symptoms with total score ranges from 0 to 32 (0 = the best quality of life; 32 = the worst quality of life with severe symptoms). ECOG assess participant's performance status on a scale of 0 to 5, where 0=fully active and 5=dead.
Time Frame: Up to 6.9 years
Population: The mITT analysis set in the Phase 2 part of this study included all participants with MET+ HCC who were randomized to study treatment. As per planned analysis, data for this outcome was analyzed only for phase 2 based on combined analysis of both FHSI-8 and ECOG.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Months | 2.2 [1.4 to 4.2] | 2.7 [0.9 to 3.7]
Statistical Analysis 1: Comparison: Phase 2: Tepotinib vs Phase 2 Sorafenib; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.8915, Log Rank; Hazard Ratio (HR) = 1.04, 90% CI [0.62 to 1.77]

20. Secondary Outcome: Phase 2: Objective Response Rate (ORR) Based on Tumor Assessment by the IRC
Description: The objective response rate (ORR) was defined as the percentage of participants who had achieved complete response (CR) or partial response (PR) as the best overall response according to radiological assessments as adjudicated by the IRC from randomization until the first occurrence of PD. CR: Complete Response (CR) defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response (PR) defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started.
Time Frame: Time from randomization until the first occurrence of PD assessed up to 6.9 years
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Percentage of participants | 10.5 [4.8 to 21.5] | 0 [0.0 to 6.8]
Statistical Analysis 1: Comparison: Phase 2: Tepotinib vs Phase 2 Sorafenib; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.0438, Cochran-Mantel-Haenszel

21. Secondary Outcome: Phase 2: Percentage of Participants With Disease Control Based on Tumor Assessment by IRC According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: Disease control was defined as CR, PR, or stable disease (SD) as the best overall response according to radiological assessments as adjudicated by the IRC from randomization until the first occurrence of PD. CR defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started. Percentage of participants with disease control were reported.
Time Frame: Time from randomization until the first occurrence of PD assessed up to 6.9 years
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Percentage of participants | 50 [37.1 to 62.9] | 21.6 [12.6 to 34.5]

22. Secondary Outcome: Phase 2: Progression-free Survival (PFS) Based on Tumor Assessment by the Investigator
Description: Progression-free survival (assessed by the Investigator) time was defined as the time in months from randomization to either first observation of radiologically confirmed progression disease by the investigator or occurrence of death due to any cause within 84 days of either randomization or the last tumor assessment. PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 mm. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from randomization to disease progression or occurrence of death due to any cause within 84 days of either randomization or the last tumor assessment, assessed up to 6.9 years
Population: as for outcome 4
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Months | 3.2 [2.7 to 5.6] | 2.8 [1.5 to 2.8]
Statistical Analysis 1: Comparison: Phase 2: Tepotinib vs Phase 2 Sorafenib; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.0496, Log Rank; Hazard Ratio (HR) = 0.59, 90% CI 2-sided [0.38 to 0.92]

23. Secondary Outcome: Phase 2: Objective Response Rate (ORR) Based on Tumor Assessment by the Investigator
Description: The objective response rate was defined as the percentage of participants who had achieved CR or PR as the best overall response according to radiological assessments as adjudicated by the investigator from randomization until the first occurrence of PD. CR defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started.
Time Frame: Time from randomization until the first occurrence of PD assessed up to 6.9 years
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Percentage of participants | 15.8 [8.4 to 27.7] | 2.7 [0.6 to 11.2]
Statistical Analysis 1: Comparison: Phase 2: Tepotinib vs Phase 2 Sorafenib; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.0527, Cochran-Mantel-Haenszel

24. Secondary Outcome: Phase 2: Percentage of Participants With Disease Control Based on Tumor Assessment by Investigator According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: as for outcome 21
Time Frame: Approximately up to 6.9 years
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: Tepotinib | Phase 2 Sorafenib
Number analyzed (Participants) | 38 | 37
Percentage of Participants | 60.5 [47.2 to 72.4] | 45.9 [33.2 to 59.2]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 30 after the last dose of study treatment, assessed up to 94 weeks (Phase 1b) and 6.9 years (Phase 2).
Description: The safety analysis set included all participants who had received any dose of the study medication.
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 1b: Tepotinib 1000 mg | Phase 2: Tepotinib | Phase 2 Sorafenib
All-Cause Mortality (participants affected / at risk) | 7/7 | 11/14 | 3/6 | 24/45 | 30/44
Serious Adverse Events (participants affected / at risk) | 2/7 | 9/14 | 4/6 | 23/45 | 12/44
Other Adverse Events (participants affected / at risk) | 7/7 | 14/14 | 6/6 | 43/45 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Tepotinib 300 mg (N=7) | Phase 1b: Tepotinib 500 mg (N=14) | Phase 1b: Tepotinib 1000 mg (N=6) | Phase 2: Tepotinib (N=45) | Phase 2 Sorafenib (N=44)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Encapsulating peritoneal sclerosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 7 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Tepotinib 300 mg (N=7) | Phase 1b: Tepotinib 500 mg (N=14) | Phase 1b: Tepotinib 1000 mg (N=6) | Phase 2: Tepotinib (N=45) | Phase 2 Sorafenib (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 2
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 4 | 0 | 9 | 5
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 6 | 1 | 11 | 9
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 7
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 3 | 3 | 11 | 4
Constipation (Gastrointestinal disorders) | 1 | 4 | 4 | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 4 | 16 | 17
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 1 | 4 | 6
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 2 | 4 | 7
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 3 | 6
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 5
Chest pain (General disorders) | 0 | 0 | 0 | 3 | 2
Fatigue (General disorders) | 1 | 3 | 2 | 12 | 13
Disease progression (General disorders) | 0 | 0 | 0 | 3 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 1 | 1 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 3 | 1
Oedema peripheral (General disorders) | 2 | 4 | 1 | 20 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 2 | 7 | 7
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 3 | 3
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 3 | 7 | 9
Amylase increased (Investigations) | 0 | 2 | 1 | 4 | 7
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 4 | 10 | 16
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 3 | 5 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 4 | 11
Blood creatinine increased (Investigations) | 1 | 0 | 3 | 7 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Creatinine renal clearance increased (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 3 | 8
Lipase increased (Investigations) | 0 | 3 | 1 | 2 | 8
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 2 | 4
Platelet count decreased (Investigations) | 0 | 0 | 1 | 7 | 7
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 3
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 9
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2 | 16 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 4 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 5 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 12 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 1 | 2 | 5
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 3
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Penile swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 11
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 11 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4 | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 12
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT01988493/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT01988493/SAP_001.pdf